CLINICAL TRIAL: NCT07251998
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Phase 2 Clinical Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of ICP-332 in Patients With Moderate to Severe Plaque Psoriasis
Brief Title: Efficacy and Safety of ICP-332 Versus Placebo in Participants With Moderate to Severe Plaque Psoriasis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICP-CL-00603
Record Dates: First submitted 2025-11-19; First posted 2025-11-26 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ICP-332 Dose A (Experimental)
  Interventions: Drug: ICP-332 Tablets
- ICP-332 Dose B (Experimental)
  Interventions: Drug: ICP-332 Tablets
- ICP-332 Dose C (Experimental)
  Interventions: Drug: ICP-332 Tablets
- ICP-332 Placebo (Placebo Comparator)
  Interventions: Other: ICP-332 Placebo Tablets

INTERVENTIONS:
Drug: ICP-332 Tablets — ICP-332 will be administered as tablet for 12 weeks
  Arms: ICP-332 Dose A
Drug: ICP-332 Tablets — ICP-332 will be administered as tablet for 12 weeks
  Arms: ICP-332 Dose B
Drug: ICP-332 Tablets — ICP-332 will be administered as tablet for 12 weeks
  Arms: ICP-332 Dose C
Other: ICP-332 Placebo Tablets — Placebo will be administered as tablet for 12 weeks
  Arms: ICP-332 Placebo

SUMMARY:
The purpose of this study is to compare the efficacy and safety of ICP-332 to placebo in participants with moderate-to-severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in this study and have signed the Informed Consent Form (ICF).
2. Male or female subjects aged ≥ 18 years and ≤ 70 years
3. A history of plaque psoriasis for ≥6 months at baseline
4. Meet the following three criteria:

   1. Psoriasis Area and Severity Index (PASI) score ≥12
   2. Static Physician's Global Assessment (sPGA) score ≥3
   3. Psoriasis affected Body Surface Area (BSA) ≥10%
5. The subject requires systemic treatment and/or phototherapy.

Exclusion Criteria:

1. Diagnosed with non-plaque psoriasis.
2. Subject had laboratory values meeting any of the protocol-specified criteria at Screening.
3. Presence of clinically serious, progressive, or uncontrolled disease.
4. Previous history of alcoholism or drug abuse (except for those who have been completely abstinent for more than 6 months before randomization).
5. Pregnant or lactating women.
6. The investigator accepts ICP-332 for any reason that the subject is not suitable for this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
The Percentage of Participants With Moderate to Severe Psoriasis Experiencing a 75% Improvement (Reduction From Baseline) in PASI Score (PASI-75 Response Rate) at Week 12 | Day 1 to Day 85

CONTACTS AND LOCATIONS:
Overall Officials: Yuling Shi, Principal Investigator — Shanghai Dermatology Hospital
Locations (1):
- Shanghai Dermatology Hospital, Shanghai, Shanghai Municipality, China